CLINICAL TRIAL: NCT04096469
Title: Intervention Program to Promote Changes in Diet and Physical Activity and to Evaluate Its Impact on Body Weight, Biomarkers of Disease and Quality of Life in Breast Cancer Survivors
Brief Title: Impact of Diet and Physical Activity Changes on Body Weight, Biomarkers and Quality of Life in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigación en Alimentación y Desarrollo A.C. (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Graciela Caire Juvera, PhD, PhD, Centro de Investigación en Alimentación y Desarrollo A.C.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 60252; 262211 (Other: Conacyt)
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Body Weight Changes; Mammographic Density; Quality of Life
Keywords: breast cancer survivors; diet; physical activity; motivational interviewing; body weight; quality of life; biomarkers
MeSH Terms: conditions — Body Weight Changes; Motor Activity; Body Weight | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: The intervention group received the motivational interviewing and the comparison group an orientation with a traditional educational approach. Both groups were followed for 8 months and the changes in the variables of interest were analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): The intervention group received a guidance regarding their diet and physical activity using the motivational interviewing strategy to improve adherence to healthy behaviors. Participants received a guide with a motivational interviewing approach, which served as the basis for the interview process. The objectives in the intervention group were to consume four vegetables and two fruits a day, seven days a week, increase fiber consumption to more than 30 g daily, reduce fat consumption to no more 20% of the total energy consumed, decrease the consumption of sugary drinks and increase protein intake. Another goal was to increase the number of steps to 4,000 additional steps to those who have already walked.
  Interventions: Behavioral: Motivational Interviewing
- Traditional Education (Active Comparator): The comparison group received a guide on medical care and nutrition with a traditional educational approach. The indication was to read and learn about the health-related topics included in the booklet that was given to them. These participants were visited in the same way as the intervention group to answer questions and monitor participation throughout the intervention.
  Interventions: Behavioral: Traditional Education

INTERVENTIONS:
Behavioral: Motivational Interviewing — The motivational interviewing strengthens the motivation and commitment to achieve a specific change through the induction and exploration of the reasons for modifying behavior. All this within an atmosphere of acceptance and compassion. It is about extracting the possible solutions to the change that is faced from the individual and his environment and not from the professional. This strategy is achieved by looking for the patient to feel motivated, and to express their problem and thus create discrepancy so that they evaluate their actions and reflect on the changes they should make.
  Other Names: Intervention group
  Arms: Motivational Interviewing
Behavioral: Traditional Education — Traditional education refers to the normal care given to breast cancer survivors. That is, they receive recommendations about their physical activity and diet but without any motivational approach.
  Other Names: Comparison group
  Arms: Traditional Education

SUMMARY:
This study is a randomized controlled clinical trial of two arms, which included 60 women survivors of breast cancer of the state of Sonora, Mexico.The intervention is for 8 months and includes home visits every 15 days for the first four months and monthly for the last four months.The objective was to evaluate the effect of a diet and physical activity intervention program using the motivational interviewing (MI) strategy compared to an orientation with a traditional educational approach to improve anthropometric variables such as body weight, fat, muscle mass and bone mineral density, as well as biomarkers of the disease such as mammographic density, telomere length, telomerase activity, DNA methylation, ceramide-1-phosphate transport protein (CPTP), vascular endothelial growth factor (VEGF), C-reactive protein (CRP), interlucin 6 (IL-6) , interlucin 8 (IL-8), tumor necrosis factor alpha (TNF-α), leptin and adiponectin. Finally, the study also aims to improve psychological variables such as quality of life, sleep quality, anxiety and optimism.

DETAILED DESCRIPTION:
The overall objective was to design and implement an intervention program to promote changes in diet and physical activity that promotes, through the focus of the motivational interview, the increase in the consumption of fruits and vegetables, the decrease in the consumption of fats and the increase in physical activity, to achieve an impact in the reduction of weight and body fat, the improvement in the biomarkers of the disease and in the quality of life in women survivors of BC.

Specific objectives

1. Determine the adherence of participants to a healthy lifestyle intervention by analyzing biological markers of dietary intake (alpha and beta carotene, as well as lipid profile) at the beginning of the study and at 4 and 8 months after initiation of the intervention.
2. Investigate the impact of the intervention on changes in weight, body mass index, body fat, muscle mass and bone mineral density of women by measuring these variables at the beginning of the study and at 4 and 8 months after intervention.
3. Examine the effect of the intervention on biomarkers of the disease: mammographic density, telomere length and telomerase activity, VEGF, DNA methylation and CPTP at baseline and 8 months.
4. To evaluate the impact of the intervention program on inflammatory markers: leptin and adiponectin, IL6, IL8, CRP and TNF-α at the beginning, 4 and 8 months after the intervention started.
5. Analyze the effect of the intervention on the alterations in sleep quality and quality of life of the women survivors of breast cancer at the beginning, 4 and 8 months after the intervention.

Study Design and Participants

This was a randomized controlled clinical trial with two groups of breast cancer survivors. In the intervention group, we used the strategy of Motivational Interviewing to promote changes in diet and physical activity; the comparison group received an orientation with a traditional educational approach. The intervention program lasted eight months. A total of 60 women from Sonora, Mexico, participated in the study. The women were selected from the State Oncology Center and through social networks. The research protocol was sent to the ethics committee of the Center for Research in Food and Development, A.C. and women signed an informed consent letter to participate in the study.

Visits and monitoring

After the recruitment, application of questionnaires and blood sampling at the first visit (baseline), the participants were randomly assigned to the intervention (n = 30) or the comparison group (n = 30). The orientation was similar in both groups and was carried out in two modalities: in person at the participant's house and by telephone. The first orientation was made within the first 15 days after the first visit (baseline) and was at the participant's home. Within a week of the first initial orientation, the participants were called by phone to continue the monitoring and orientation process. During the first four months, the orientation was every fifteen days, and combined the visits to the participant's house with phone calls. During the next four months, the orientation took place once a month and at the participant's house.

Intervention program for changes in lifestyle

Guidance on lifestyle changes in the intervention group was carried out using the motivational interviewing approach and was conducted by trained personnel for that purpose. The dietary intervention was designed to promote the increase in plasma carotene levels, due to the increase in the consumption of fruits and vegetables. The intervention also promoted the improvement of the lipid profile (due to the decrease in fat consumption) and the control or reduction of body weight.

The diet and physical activity components of the lifestyle change program were progressive, and we managed individualized interventions. Both the diet and the physical activity regimen could be adjusted to any unexpected situation (e.g., Decrease in the number of steps due to stomach problems or ankle sprains) during the entire participation period.

The dietary goals contemplated to reach a consumption of 20% of the total energy coming from fats, the consumption of 6 or more servings of fruits / vegetables a day and the promotion of a healthy body weight, to increase fiber consumption to a greater than 30 grams daily, decrease the consumption of sugary drinks and increase the consumption of protein. The emphasis on dietary fat restriction helped to achieve other dietary goals, such as increased consumption of vegetables and fruits, increased fiber consumption, and mild to moderate body weight loss. To reach the goal of having a fat intake in the diet of 20% of the total energy consumed, a goal of grams of fat was established for each participant.

The component of physical activity consisted of a moderately low aerobic regime with the aim of gradually increasing the number of steps per week, in order to be able to walk at least 4000 steps (in addition to those that are already routine) per day or 28,000 steps per week. In addition, participants were encouraged to reduce sedentary time, by performing simple exercises while sitting and stretching exercises, among others.

The educational materials covered different topics such as knowing how to read and interpret the labels on food, recommendations for buying food, recommendations for eating out and others. The visits and orientation calls included a brief assessment of the food consumed and the physical activity performed the previous day, as well as a review of the list of weekly behavior goals and lifestyle journals, which helped the counselor to assess adherence to lifestyle goals and provide specific encouragement and feedback to the participant. Lifestyle journals were used to assess the intake of fat grams as well as daily steps to assess adherence and identify specific barriers to compliance with behavioral goals.

Comparison group

This group received a notebook that included general health information. As with the intervention group, they were provided with a pedometer and common literature on recommendations to stay physically active. Participants in this group were not asked to record their diet or physical activity, and guidance was provided monthly during the 8-month intervention.

Collection of information

The collection of the information was carried out in the two groups. The sociodemographic and health data of the participants were obtained in the first visit. The anthropometric and body composition measurements, as well as the application of questionnaires on sleep quality and quality of life were carried out at the first visit (day 1), 4 and 8 months after the intervention as well the dietary evaluation. The blood samples for the analysis of carotenoids, lipid profile, , VEGF, DNA methylation, and proinflammatory markers were taken on the first day, at 4 and 8 months. The mammographic density analysis, telomere length, and telomerase activity were carried out at the beginning of the study and at 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 with a diagnosis of stage II-IV invasive breast cancer
* Have at least 6 weeks and no more than 2 years of completing your therapy at the time of recruitment
* Do not present metastasis
* Not having a special diet or rigorous physical activity
* Not suffer any chronic illness or physical limitation
* Not have depression problems
* Sign the informed consent letter

Exclusion Criteria

* Have restrictions for physical activity
* Strict diet or be a vegetarian
* Body mass index below 18
* Having undergone surgery to lose weight
* Having excision in both breasts or having implants

Ages: 18 Years to 73 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | baseline, at four months and eight months
  Change in body weight in kilograms
Change in Breast Density | baseline and at eight months
  Change in the amount of dense tissue compared to the amount of fatty tissue in the breast on a mammogram reported in percentage
Change in Quality life | baseline, at four months and eight months
  Change in score of the scale of the Quality of Life Patient/Cancer Survivor Version. questionnaire carried out by Ferrell et al., (2012). This questionnaire analyzes the dimensions of physical, emotional, social, and spiritual well-being through a Likert scale. The minimum score to be obtained is 42 and the maximum score is 210 points, where the higher the score, the better the quality of life and the lower the score, the worse the quality of life.
Change in Sleep Quality | baseline, at four months and eight months
  Change in score of the scale of the Pittsburgh Sleep Quality Index. This questionnaire uses a Likert-type scale and provides an overall score of the quality of sleep in a range of 0 to 21, where the highest score refers to greater difficulties in all areas of sleep and a lower score gives a better sleep quality
Change in telomere length | baseline and at eight months
  Absolute telomere length (kilobase pair) (kbp)
Change in Bone Mineral Density | baseline, at four months and eight months
  The amount of bone mineral in bone tissue in g/cm2

SECONDARY OUTCOMES:
Change in the activity of telomerase | baseline and at eight months
  absorbance in nanometers
Change in C-reactive protein levels | baseline and at eight months
  miligramos por litro (mg/L)
Change in interleukin 6 levels | baseline and at eight months
  picograms per milliliter pfg / mL
Change in interleukin 8 levels | baseline and at eight months
  picograms per milliliter (pg / mL)
Change in levels of tumor necrosis factor alpha | baseline and at eight months
  picograms per milliliter (pg / mL)
Change in vascular endothelial growth factor levels | baseline and at eight months
  Picograms per milliliter (pg / mL)
Change in leptin levels | baseline and at eight months
  nanograms per milliliter (ng / mL).
Change in adiponectin levels | baseline and at eight months
  nanograms per milliliter (ng / mL).
Change in the percentage of fat mass | baseline, at four months and eight months
  Change in percentage
Change in percentage of muscle mass | baseline, at four months and eight months
  Change in percentage
change in the optimism scale | baseline, at four months and eight months
  The Revised Vital Orientation Test (LOT-R) was used, which is made up of a total of 10 items with a Likert response with five response options (from 0 = "strongly disagree" to 4 = "strongly agree "). The higher the level of optimism, the higher the level of optimism.
change in the anxiety scale | baseline, at four months and eight months
  The State-Trait Anxiety Inventory, STAI was used. This questionnaire has twenty items for each of the subscales that are state anxiety and trait anxiety, with an alternative Likert response scale (from 0 = "nothing" to 3 = "a lot" for state anxiety and for trait anxiety of 0 = "Almost never" to 3 = "almost always"). Totals range from 0 to 60 for each subscale, a higher score reflects higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Graciela Caire Juvera, PhD, Principal Investigator — CIAD
Locations (1):
- Centro de Investigación en Alimentación y Desarrollo, Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: No
Actually there is no plan to share IPD to other researchers